CLINICAL TRIAL: NCT03230266
Title: Determination of the Root Causes of Obstructions of Catheters in Patients With Type 1 Diabetes Treated by Insulin Implanted Pumps
Brief Title: Root Cause Determination of Catheter Obstructions
Acronym: CATS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9802
Record Dates: First submitted 2017-05-17; First posted 2017-07-26 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collection (Other): collection of biological and device samples
  Interventions: Procedure: Collection of intra-peritoneal catheters for insulin infusion

INTERVENTIONS:
Procedure: Collection of intra-peritoneal catheters for insulin infusion — Collection of intra-peritoneal catheters for insulin infusion

SUMMARY:
During this study, the investigators will perform a collection of biological and device samples (blood, catheters, insulin) in order to investigate the causes of catheter obstructions in patients with type 1 diabetes treated by implanted insulin pumps using intra-peritoneal delivery.

This multi-centre study is interventional with minimal constraints. After an inclusion visit, blood samples and an insulin sample from pump reservoir will be collected. During the following year, if a peritoneal catheter is blocked or changed, the explanted catheter and new blood and insulin samples will be collected for examination of the catheter obstruction and search for patient- or insulin-related reasons for obstructions.

In this study, 140 patients will be investigated.

DETAILED DESCRIPTION:
In patients with type 1 diabetes treated by implanted pumps using intra-peritoneal delivery, the incidence of peritoneal catheter obstructions is close to 12 per 100 patient-years. Variability of occurrence is however important between patients. Fibrin, aggregates of insulin and fibrotic tissue have been found inside the catheter lumen at peritoneal tip or forming a capsule around the catheter. This study will investigate with more precision the nature of catheter blockages and look for potential causes of these obstructions such as stability of insulin in the pump reservoir, immune reactions against insulin or catheter components in patient plasma, prothrombotic factors in patient blood. Blood samples and insulin from pump reservoir will be collected at baseline (inclusion). During the following one year period, each catheter presenting an obstruction or needing a change associated with pump change will be collected and explored. Blood and insulin samples will be collected again for comparison with initial samples. Investigations will be performed in collaboration with Pr Burgess' team at the School of Pharmacy of the University of Connecticut. From obtained results, models replicating the conditions of obstruction will be elaborated and tested in rodents at the University of Connecticut. Solutions will be proposed to reduce the occurrence of obstruction of peritoneal catheters as an outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Collection of catheters for intra-peritoneal insulin infusion from implanted pumps presenting obstructions or not

Exclusion Criteria:

-

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Collection of catheters for intra-peritoneal insulin infusion from implanted pumps presenting obstructions or not : collection of biological and device samples (blood, catheters, insulin) | one day
  collection of biological and device samples (blood, catheters, insulin) the explanted catheter and new blood and insulin samples will be collected for examination of the catheter obstruction and search for patient- or insulin-related reasons for obstructions.

SECONDARY OUTCOMES:
Associated conditions related to the patient and to infused insulin | one day
  Our study will investigate with more precision the nature of catheter blockages and look for potential causes of these obstructions such as stability of insulin in the pump reservoir, immune reactions against insulin or catheter components in patient plasma, prothrombotic factors in patient blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided